CLINICAL TRIAL: NCT06101498
Title: The Effect of Peroperative Fluid Management Strategy on Postoperative Renal Functions in Major Gyneco-oncological Surgeries
Brief Title: Peroperative Fluid Management in Major Gynecological Cancer Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Duygu Akyol, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023.478
Record Dates: First submitted 2023-10-17; First posted 2023-10-26 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Fluid Overload; Fluid Loss; Perioperative/Postoperative Complications; Acute Kidney Injury
Keywords: akut kidney injury; goal directed fluid therapy; peroperative fluid management; conventional fluid therapy
MeSH Terms: conditions — Edema; Postoperative Complications; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional fluid therapy (Experimental): Patients who received conventional fluid therapy
  Interventions: Diagnostic Test: Akut kidnet injury(AKI)
- Non invaziv goal directed therapy (Experimental): Patients who received non invaziv goal directed therapy
  Interventions: Diagnostic Test: Akut kidnet injury(AKI)
- Minimal invaziv goal directed therapy (Experimental): Patients who received minimal invaziv goal directed therapy
  Interventions: Diagnostic Test: Akut kidnet injury(AKI)

INTERVENTIONS:
Diagnostic Test: Akut kidnet injury(AKI) — postoperative 24 hours
  Other Names: AKI developing in the patient group receiving conventional treatment; AKI developing in the patient group receiving non invaziv goal directed therapy; AKI developing in the patient group receiving minimal invaziv goal directed therapy

SUMMARY:
The aim of this study is to evaluate the effect of perioperative fluid management on postoperative kidney damage in gynecological cancer surgeries.

The main question[s] it aims to answer are:

Does fluid management applied with different hemodynamic monitoring methods affect the risk of postoperative AKI? In our clinic, three different fluid management strategies are applied depending on the anesthetist experience. Acute kidney injury will be evaluated according to the postoperative AKIN classification of conventional fluid therapy and targeted fluid therapy with noninvasive or minimally invasive monitoring.

DETAILED DESCRIPTION:
Our study was designed as a retrospective study. The files of patients over the age of 18 who underwent open abdominal surgery due to ASAII and III gynecological malignancy will be examined retrospectively. Patients who cannot be monitored peroperatively and who undergo HIPEC will be excluded from the study. Patients will be divided into 3 groups according to the fluid management strategy and the hemodynamic monitoring used: Group 1: patients receiving conventional fluid therapy; Group 2: patients receiving targeted fluid therapy with noninvasive monitoring; Group 3: patients receiving targeted fluid therapy with minimally invasive monitoring.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* ASA II-III
* Those with normal renal function

Exclusion Criteria:

* Patients in renal insufficiency
* Patients with perioperative renal, ureter & bladder invasion
* Patients in whom perioperative urine monitoring cannot be performed
* Patients undergoing HIPEC
* Patients with missing data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of acute kidney injury | Change from preoperative to postoperative day 1(POD1)creatinine values(mg/dl)
  Our primary aim was to evaluate the postoperative day(POD1 ) creatinine values(mg/dl)

SECONDARY OUTCOMES:
Peroperative fluid amounts | during the operation period
  The seconder aim to investigate the amount of fluid used peroperatively

OTHER OUTCOMES:
The intensive care unit admission | posoperatively up to 1 months
  The other aim to investigate the intensive care unit admission
Length of stay | postoperative 30 days
  The other aim to evaluate the duration of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Akyol, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Basaksehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yildiz GO, Hergunsel GO, Sertcakacilar G, Akyol D, Karakas S, Cukurova Z. Perioperative goal-directed fluid management using noninvasive hemodynamic monitoring in gynecologic oncology. Braz J Anesthesiol. 2022 May-Jun;72(3):322-330. doi: 10.1016/j.bjane.2021.12.012. Epub 2022 Feb 1. PMID 35121063
- [Result] Yu J, Che L, Zhu A, Xu L, Huang Y. Goal-Directed Intraoperative Fluid Therapy Benefits Patients Undergoing Major Gynecologic Oncology Surgery: A Controlled Before-and-After Study. Front Oncol. 2022 Apr 6;12:833273. doi: 10.3389/fonc.2022.833273. eCollection 2022. PMID 35463383
- [Result] Russo A, Aceto P, Grieco DL, Anzellotti GM, Perilli V, Costantini B, Romano B, Scambia G, Sollazzi L, Antonelli M. Goal-directed hemodynamic management in patients undergoing primary debulking gynaecological surgery: A matched-controlled precision medicine study. Gynecol Oncol. 2018 Nov;151(2):299-305. doi: 10.1016/j.ygyno.2018.08.034. Epub 2018 Sep 7. PMID 30201234
- [Result] Hasselgren E, Hertzberg D, Camderman T, Bjorne H, Salehi S. Perioperative fluid balance and major postoperative complications in surgery for advanced epithelial ovarian cancer. Gynecol Oncol. 2021 May;161(2):402-407. doi: 10.1016/j.ygyno.2021.02.034. Epub 2021 Mar 12. PMID 33715894
- [Result] McKenny M, Conroy P, Wong A, Farren M, Gleeson N, Walsh C, O'Malley C, Dowd N. A randomised prospective trial of intra-operative oesophageal Doppler-guided fluid administration in major gynaecological surgery. Anaesthesia. 2013 Dec;68(12):1224-31. doi: 10.1111/anae.12355. Epub 2013 Sep 30. PMID 24116747